CLINICAL TRIAL: NCT03115021
Title: Neurophysiological Effects of tPCS and tDCS on Patients With Disorders of Consciousness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Aurore Thibaut, Investigator, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016P001840
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Disorders of Consciousness
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active tPCS / Sham tDCS (Experimental): All subject will receive active tPCS and sham tDCS for 20 minutes simultaneously.
  Interventions: Device: Active tPCS; Device: Sham tDCS
- Sham tPCS / Active tDCS (Experimental): All subject will receive sham tPCS and active tDCS for 20 minutes simultaneously.
  Interventions: Device: Active tDCS; Device: Sham tPCS
- Sham tPCS / Sham tDCS (Experimental): All subject will receive sham tPCS and sham tDCS for 20 minutes simultaneously.
  Interventions: Device: Sham tPCS; Device: Sham tDCS

INTERVENTIONS:
Device: Active tPCS — A current intensity of 2na and a stimulation frequency range of 6-10 Hz will be used with a peri-auricular ear-clip electrode montage for 20 minutes.
  Arms: Active tPCS / Sham tDCS
Device: Active tDCS — A current intensity of 2mA will be used for 20minutes. The electrodes that will be used will be standard sponge electrodes. The anode will be place over the left prefrontal cortex and the cathode over the right supraorbitofrontal area.
  Arms: Sham tPCS / Active tDCS
Device: Sham tPCS — Sham tPCS will consist of applying the same parameters as for active but the corresponding device will be turned off after 30 seconds as to simulate the initial sensation of the active current. A current of 2mA will still be used (but turned off after 30 sec). The electrodes that will be used will be the same as for the active tPCS condition and the electrodes placement as well.
  Arms: Sham tPCS / Active tDCS; Sham tPCS / Sham tDCS
Device: Sham tDCS — Sham tDCS will consist of applying the same parameters as for active but the corresponding device will be turned off after 30 seconds as to simulate the initial sensation of the active current. A current of 2mA will still be used (but turned off after 30 sec). The electrodes that will be used will be the same as for the active tDCS condition and the electrodes placement as well.
  Arms: Active tPCS / Sham tDCS; Sham tPCS / Sham tDCS

SUMMARY:
This study aims at comparing the effects of transcranial direct current stimulation and transcranial pulsed current stimulation on neurophysiological outcomes on patients with disorders of consciousness. This study also aims to evaluate the effects of these techniques on patients' level of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English or French
* Legally authorized surrogate available to provide informed consent
* History of non-traumatic brain injury with loss of consciousness caused by stroke, cerebral hemorrhage, hypoxic ischemic insult, metabolic disorder or infection.
* Has been followed clinically on the CRS-R for a minimum two weeks and has undergone a minimum of 4 assessments with the CRS-R.
* Serial CRS-R scores show at least one subscale on which there is no behavioral sign of conscious awareness (ie, command following, visual fixation or pursuit, object localization or recognition, localization to noxious stimulation, object manipulation, automatic motor responses, functional object use, discernable speech, discernable yes no communication, based on clinically obtained scores contained in the medical record).
* CRS-R screening examination completed by research staff confirms the absence of a behavioral sign of consciousness on a least one CRS-R subscale.
* Medically stable (i.e., no systemic illness or disease) and capable of independent ventilation

Exclusion Criteria:

* History of developmental, neurologic, or major psychiatric disorder resulting in functional disability up to time of enrollment.
* Evidence or surrogate report of uncontrolled seizure disorder
* Metallic brain implant or implanted electronic brain medical devices or pacemaker
* Subjects with craniectomy
* History of cranioplasty in the frontal region or recent cranioplasty that has not yet fully healed
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Signal coherence and EEG power as measured by Quantitative electroencephalographic analysis (qEEG) | It will be measured over the course of about 3 weeks
  EEG measures cortical electrical activity and examines the dynamic changes.

SECONDARY OUTCOMES:
Coma Recovery Scale Revised (CRS-R) | It will be measured over the course of about 3 weeks
  The CRS-R is a standard clinical protocol used to assess patients' level of consciousness. This test measures the level of response to sensory stimulation, ability to understand language and to communicate.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Liege, Liège, Belgium